CLINICAL TRIAL: NCT04621747
Title: Trial Investigating the Characteristics of Knismesis - a Lever to Explore Allodynia in Neuropathic Pain
Acronym: TICKLE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: NEURO-DOL (UMR 1107 INSERM / UCA) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RBHP 2020 DUALE
Record Dates: First submitted 2020-11-02; First posted 2020-11-09 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-12

CONDITIONS: Healthy
Keywords: Neurophysiology; Psychophysics; Sensory thresholds; Neurons; Pain, neuropathic
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): healthy volunteers aged 18-35, balanced sex ratio, all of them undergoing the same battery of psychophysical explorations.
  Interventions: Other: Battery of neurophysiological explorations

INTERVENTIONS:
Other: Battery of neurophysiological explorations — Visit 1: Biometry collection: gender, age, weight, height, eye colour.
  * Questionnaires : the State and Trait Anxiety Inventory and the Pain Sensitivity
  * Threshold of unpleasant light brightness, mechanical sensitivity threshold (von Frey hair).
  * Training to estimate unpleasantness Under nociceptive and tickling stimuli, to use the handgrip.
  * Mechanical pain threshold (electronic von Frey), heat pain threshold (Medoc Pathway).
  * 48 stimulations applied to the back skin, following a predetermined plan with 12 different pathways, imbricated with 4 different speeds of movement.
  Visit 2 (1 to 8 days later) :
  * 42 stimulations applied to the back skin, to test the effect of stimulation intensity, the side of application, continuity break of the contact, and distraction by other cutaneous stimuli. The stimuli will follow the best paradigm as identified at the previous visit.
  * 12 stimulations applied to forearm, cheeks, lower limbs, also testing the effect of hairiness.

SUMMARY:
Also known as a "moving itch", knismesis is a mildly annoying sensation caused by a light movement on the skin, such as from a crawling insect. Its underlying mechanism rely on spatial summation, i.e. amplification of the signal due to summation of stimulated fields, like it is for dynamic allodynia in neuropathic pain. This physiological study aims at determining the physical factors of the cutaneous stimulation inducing knismesis as well as the effect of confounding factors. The main area of exploration will be the back, because of its size and the possibility to blind the participant. The information collected, along with animal data in surrogate models, would help to better understand neuropathic pain in the future.

DETAILED DESCRIPTION:
This is a physiological proof-of-concept, also aiming to validate a functional exploration model in healthy volunteers. Each participant will undergo a battery if psychometric then psychophysics tests, presented sequentially. However, most of the main study tests (knismesis) will be admistered in a random order (crossover). The primary endpoint is to characterise, in the healthy human, the physical determinants of the cutaneous stimulation inducing knismesis: length of the pathway, speed, direction, intensity, continuity break of the contact, hairiness, body site, or distraction by other cutaneous stimuli. The secondary endpoint is to study the relationship between the individual sensitivity to spatial summation (knismesis) and other individual sensitivities or profiles.

ELIGIBILITY:
Inclusion Criteria:

- Ability to answer French questionnaires.

· BMI between 19 and 30 kg/m2 at inclusion.

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Natural intolerance to tickling.
* Any cutaneous, ocular or neurological disease contraindicating the psychophysical tests.
* Any disease or medical history that could expose the subject to unacceptable risk during the study.
* Any medication intake within 7 days before testing.
* History of drug or alcohol abuse.
* Involvement in another concomitant research protocol.
* Major dorsal hairiness.
* Inability to undergo the tests.
* Legal protection.
* Concomitant involvement in another clinical research.
* Refusal to participate.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-11-23 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Intensity of annoying sensation | Day 1
  After training, the annoying sensation is expressed by the subject through a handgrip dynamometer (Biopac systems). The signal will be treated and converted into area-under-curve response (Dualé C et al., Reg Anesth Pain Med 2011; 36:110-115).
Intensity of annoying sensation | Day 8
  After training, the annoying sensation is expressed by the subject through a handgrip dynamometer (Biopac systems). The signal will be treated and converted into area-under-curve response (Dualé C et al., Reg Anesth Pain Med 2011; 36:110-115).

SECONDARY OUTCOMES:
Muscular aversive response. | Day 1, Day 8
  The muscular aversive response will be assessed by surface electromyography through paraspinal contact electrodes (Biopac systems).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Clermont Ferrand, Clermont-Ferrand, Auvergne, France